CLINICAL TRIAL: NCT06539585
Title: Scanning the Meiotic Spindle in Assisted Reproductive Techniques to Assess Oocyte Quality (SMART Study)
Brief Title: Scanning the Meiotic Spindle in Assisted Reproductive Techniques to Assess Oocyte Quality
Acronym: SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Czech Academy of Sciences (Other); Czech Technical University in Prague (Other); General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Jaromír Mašata, Leading doctor of the Center of Urogynecology and Pelvic Recontructive Surgery, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MW24-08-00048
Record Dates: First submitted 2024-07-23; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Infertility; Infertility, Male; Infertility, Female
Keywords: infertility; human oocyte; IVF; meiotic spindle; ICSI; sperm count
MeSH Terms: conditions — Infertility; Infertility, Male; Infertility, Female | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard ICSI without meiotic spindle imaging. (Active Comparator): A control group of patients who underwent a standard IVF cycle without microscopy of the meiotic spindle. In this control group of patients, ICSI fertilization will be performed 5-6 hours after oocyte collection.
  ICSI will be performed according to standard protocol [6]. The oocytes will be cultivated individually, and their order preserved, so that the other outcomes (data from timelapse, clinical results) can be associated with individual oocytes. Fertilization after ICSI will be defined as the presence of two pronuclei and 2 polar body. Embryos will be cultivated for 122-144 h.
  Interventions: Procedure: ICSI
- Meiotic spindle imaging followed by standard ICSI. (Active Comparator): MS evaluation will take place in pre-prepared glass-bottomed dishes with about 5μl medium with the HEPES buffer covered with paraffin oil, put to heat one hour before use. The oocyte will be rotated using a needle so that PB and MS are both well visible, and photographs will be taken using optical microscope. The MS status and the angle (α) between MS and PB will be obtained 3-4 hours after oocyte pick-up (OPU). At the same time, the polarized-light microscopy image will be acquired (polarized light microscopy at ×100 magnification. ICSI will be performed typically 2-3 h after the polarization microscopy evaluation, i.e., 5-6 h after OPU.
  ICSI will be performed according to standard protocol [6]. Fertilization after ICSI will be defined as the presence of two pronuclei and 2 polar body. Embryos will be cultivated for 122-144 h.
  Interventions: Procedure: Meiotic spindle status observation in polarized light; Procedure: ICSI
- MS imaging and ICSI fertilization according MS status. (Active Comparator): Oocytes with MS evaluation will be fertilized according to MS status either 5-6 hours after ovum pick-up (OPU) or 7-8 hours after OPU. MS evaluation will take place in pre-prepared glass-bottomed dishes. The MS status and the angle (α) between MS and PB will be obtained 3-4 hours after oocyte pick-up (OPU). At the same time, the polarized-light microscopy image will be acquired (polarized light microscopy at ×100 magnification. For oocytes with PB/MS in close proximity (angle between PB and MS < 5◦) or MS not visible ICSI will be performed 4-5 h after the polarization microscopy evaluation, i.e., 7-8 h after OPU (these oocytes are supposed to be not fully mature). For oocytes with MS clearly visible and PB/MS not in close proximity (angle between PB and MS > 5◦) ICSI will be performed typically 2-3 h after the polarization microscopy evaluation, i.e., 5-6 h after OPU.
  ICSI will be performed according to standard protocol [6].
  Interventions: Procedure: Meiotic spindle status observation in polarized light; Procedure: ICSI

INTERVENTIONS:
Procedure: Meiotic spindle status observation in polarized light — In patients older than 35 years and younger than 40 years, we will use a microscope with a polarizing filter to evaluate the position of meiotic spindles and polar bodies in oocytes collected from patients who were indicated for IVF and ICSI. Using an optical microscope with a Nikon CEE GmbH polarizing filter, the angle between PB and MS together with MS visibility will be determined.
  Arms: MS imaging and ICSI fertilization according MS status.; Meiotic spindle imaging followed by standard ICSI.
Procedure: ICSI — ICSI will be performed according to standard protocol using ICSI/holding micropipettes (#002-5-30/#001-120-30, Microtech IVF, Czech Republic), polyvinylpyrrolidone (ICSI™, Vitrolife, Sweden), and Eppendorf (Hamburg, Germany) micromanipulation system equipped with thermoplate (Tokaohit, Japan). The oocytes will be cultivated individually, and their order preserved, so that the other outcomes (data from timelapse, clinical results) can be associated with individual oocytes. Oocytes will be denuded (HYASE-10X™, Vitrolife, Sweden) after OPU, and the maturation stage will be examined.

SUMMARY:
The assisted reproduction success rate is affected by several factors including the age of the women, oocyte quality and maturation state, as well as sperm quality. Imaging of the meiotic spindle may be crucial for determining the oocyte maturation and the optimal time of oocyte fertilization by intracytoplasmic sperm injection (ICSI). A new accurate and non-invasive method for selecting quality maturated oocytes based on meiotic spindle imaging is for women over 35 years of age will be introduced. The evaluation of efficiency using meiotic spindle visibility in polarized light and its relative position to the polar body as indicator of oocyte maturity will be monitored and the optimal time for ICSI will be defined.

DETAILED DESCRIPTION:
One of the main strategies of infertility treatment is in vitro fertilization (IVF) . The IVF success rate is affected by several key factors including the age of the women, oocyte quality and maturation state, as well as sperm quality. Several authors have suggested that the presence, position and retardance of the optically birefringent meiotic spindle (MS) are related to oocyte developmental competence, affecting the quality of fertilization and embryo development. Oocytes with normal spindle morphology are significantly more likely to produce euploid embryos compared with oocytes with meiotic spindles that are not visible or abnormal. Adjusting the timing of intracytoplasmic sperm injection (ICSI) based on MS morphology has also been proposed. It was shown that adjusting the time of ICSI based on the position of the MS with respect to the polar body (PB) increases the probability of successful fertilization for women over 35 years of age. For the oocytes of patients over 35 years of age, the longer incubation time enabled a greater number of oocytes to become fully mature (MII phase) and prepared for ICSI. In this situation, the MS status was an important indicator of oocyte immaturity.

Patient will be randomized into three groups using Research Electronic Data Capture (REDCap): group 1, standard ICSI without MS imaging; group 2, MS imaging followed by standard ICSI, group 3, MS imaging and ICSI fertilization according MS status. Oocytes from group 3 patients with MS evaluation will be fertilized according to MS status either 5-6 hours after ovum pick-up (OPU) or 7-8 hours after OPU. Oocytes without MS evaluation will all fertilized 5-6 hours after OPU. MS evaluation will take place in pre-prepared glass-bottomed dishes with about 5μl medium with the HEPES buffer covered with paraffin oil, put to heat one hour before use. The oocyte will be rotated using a needle so that Polar Body (PB) and MS are both well visible, and photographs will be taken using optical microscope. The MS status and the angle (α) between MS and PB will be obtained 3-4 hours after oocyte pick-up (OPU). At the same time, the polarized-light microscopy image will be acquired (polarized light microscopy at ×100 magnification. Specially, for oocytes from group 3 patients with PB/MS in close proximity (angle between PB and MS < 5◦) or MS not visible will be predicted as immature oocytes. For these oocytes, ICSI will be performed 4-5 h after the polarization microscopy evaluation, i.e., 7-8 h after OPU. For oocytes with MS clearly visible and PB/MS not in close proximity (angle between PB and MS > 5◦) ICSI will be performed typically 2-3 h after the polarization microscopy evaluation, i.e., 5-6 h after OPU, as for patients from 1 and 2 groups. ICSI will be performed according to standard protocol using ICSI/holding micropipettes (Microtech IVF, Czech Republic), polyvinylpyrrolidone (ICSI™, Vitrolife, Sweden), and Eppendorf (Hamburg, Germany) micromanipulation system equipped with thermoplate (Tokaohit, Japan). The oocytes will be cultivated individually, and their order preserved, so that the other outcomes (data from timelapse, clinical results) can be associated with individual oocytes. We will also monitor the time from the human chorionic gonadotropin (hCG) administration to the completion of the actual fertilization. The oocytes will be denuded (HYASE-10X™, Vitrolife, Sweden) after OPU, and the maturation stage will be examined. Germinal Vesicle (GV) stage oocyte will not be included. Oocytes and embryos in time-lapse incubator from the Japanese manufacturer Astec will be cultivated in a timelapse dish Origio, Denmark Sage 1-Step™, Origio, Denmark under paraffin oil (OVOIL™, VITROLIFE, Sweden) at 37.0 °C, 6% CO2 and 5%O2. Fertilization after ICSI will be defined as the presence of two pronuclei and 2 polar body 16-20 h post ICSI. Embryos will be cultivated for 122-144 h.

Pilot findings will be confirmed in a randomized control trial, i.e. to the efficiency of using MS visibility and relative position to the polar body as indicators of oocyte maturation in order to optimize ICSI timing will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent ICSI;
* Spermiogram containing at least 0.5 mil/ml sperms;
* Morphlogy: normal morphology >1%;
* Stimulated cycles

Exclusion Criteria:

* Age under 35 years or over 40;
* Native cycles;
* Severe uterine abnormalities (submucosal fibroid, fibroid ≥5cm, uterine septum, endometrial polyps, uterus duplex)

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 164 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate of patients whose ICSI time was established according to MS state | 6-8 weeks
  The percentage of all attempts that leads to pregnancy of patients whose ICSI fertilization was done according MS status. Meiotic spindle visibility in polarized light and its relative position to the polar body as indicator of oocyte maturity will be monitored and the optimal time for ICSI will be defined.

SECONDARY OUTCOMES:
clinical pregnancy rate of patients whose ICSI time was not established according to measured MS state | 6-8 weeks
  The percentage of all attempts that leads to pregnancy of patients whose ICSI fertilization was not done according MS status. But the meiotic spindle visibility in polarized light and its relative position to the polar body was measured.

OTHER OUTCOMES:
Clinical pregnancy rate of patients with standard ICSI time | 6-8 weeks
  The percentage of all attempts that leads to pregnancy of patients whose ICSI was standard.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital in Prague, Prague, Czechia

REFERENCES:
- [Background] van Loendersloot LL, van Wely M, Limpens J, Bossuyt PM, Repping S, van der Veen F. Predictive factors in in vitro fertilization (IVF): a systematic review and meta-analysis. Hum Reprod Update. 2010 Nov-Dec;16(6):577-89. doi: 10.1093/humupd/dmq015. Epub 2010 Jun 25. PMID 20581128
- [Background] Wu B, Shi J, Zhao W, Lu S, Silva M, Gelety TJ. Understanding reproducibility of human IVF traits to predict next IVF cycle outcome. J Assist Reprod Genet. 2014 Oct;31(10):1323-30. doi: 10.1007/s10815-014-0288-y. Epub 2014 Aug 15. PMID 25119191
- [Background] Hanevik HI, Hessen DO. IVF and human evolution. Hum Reprod Update. 2022 Jun 30;28(4):457-479. doi: 10.1093/humupd/dmac014. PMID 35355060
- [Background] Rienzi L, Ubaldi F, Martinez F, Iacobelli M, Minasi MG, Ferrero S, Tesarik J, Greco E. Relationship between meiotic spindle location with regard to the polar body position and oocyte developmental potential after ICSI. Hum Reprod. 2003 Jun;18(6):1289-93. doi: 10.1093/humrep/deg274. PMID 12773461
- [Background] Innocenti F, Fiorentino G, Cimadomo D, Soscia D, Garagna S, Rienzi L, Ubaldi FM, Zuccotti M; SIERR. Maternal effect factors that contribute to oocytes developmental competence: an update. J Assist Reprod Genet. 2022 Apr;39(4):861-871. doi: 10.1007/s10815-022-02434-y. Epub 2022 Feb 15. PMID 35165782
- [Background] Rienzi L, Vajta G, Ubaldi F. Predictive value of oocyte morphology in human IVF: a systematic review of the literature. Hum Reprod Update. 2011 Jan-Feb;17(1):34-45. doi: 10.1093/humupd/dmq029. Epub 2010 Jul 16. PMID 20639518
- [Result] Tepla O, Topurko Z, Jirsova S, Moosova M, Fajmonova E, Cabela R, Komrskova K, Kratochvilova I, Masata J. Timing of ICSI with Respect to Meiotic Spindle Status. Int J Mol Sci. 2022 Dec 21;24(1):105. doi: 10.3390/ijms24010105. PMID 36613547